CLINICAL TRIAL: NCT05704231
Title: The Effect of Telephone-Assisted Smoking Cessation Program on Self-Efficacy, Smoking Behavior, Tumor Recurrence and Progression in Patients Diagnosed With Non-Muscle Invasive Bladder Cancer
Brief Title: The Effect of Telephone-Assisted Smoking Cessation Program in Patients Diagnosed With Non-Muscle Invasive Bladder Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: iremozdemir
Record Dates: First submitted 2022-12-22; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Non-Muscle Invasive Bladder Cancer; Self Efficacy; Smoking Behaviors; Tumor Recurrence; Progression, Disease
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Smoking; Recurrence; Disease Progression

STUDY DESIGN:
Intervention Model Description: This study is a parallel group randomized controlled study.
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention Group (Experimental): Motivational Interviewing with WhatsApp video call The individuals in the intervention group will be given a smoking cessation education and motivational interview with a WhatsApp video call for 3 months. The motivational interview will be applied every two weeks, 6 times in total. Self-efficacy scale and smoking behavior scale will be administered again at 3, 6 and 12 months after the intervention. tumor recurrence and progression will be checked by cystoscopy at 3rd and 12th months
  Interventions: Behavioral: Behavioral: Motivational Interviewing with WhatsApp video call
- No Intervention: Control Group (No Intervention): the control group received the routine care/education provided in the hospital. Self-efficacy scale and smoking behavior scale will be administered again at 3, 6 and 12 months after the routin hospital care. Both intervention and control groups' tumor recurrence and progression will be checked by cystoscopy at the 3rd and 12th months

INTERVENTIONS:
Behavioral: Behavioral: Motivational Interviewing with WhatsApp video call — The intervention group will be given a motivational interview with a WhatsApp video call for 3 months. Motivational interviews will be applied every two weeks, 6 times in total.
  Arms: Experimental: Intervention Group

SUMMARY:
This study will be carried out to examine the effect of telephone-assisted smoking cessation program on self-efficacy, smoking behavior, tumor recurrence and progression in patients with non-muscle invasive bladder cancer.

DETAILED DESCRIPTION:
This study will be conducted to examine the effect of a telephone-assisted smoking cessation program (3 months) on self-efficacy, smoking behavior, tumor recurrence and progression for chronic disease management in patients diagnosed with non-muscle invasive bladder cancer. After 3 months of motivational interviewing was applied to the experimental group, the scales will be applied in the 3rd, 6th and 12th months. The cystoscopy will be performed at 3 and 12 months for tumor recurrence and progression

ELIGIBILITY:
Inclusion Criteria:

* Being 21 years or older
* First-time diagnosis of non-muscle invasive bladder cancer (patients with pTa urothelial cancer)
* Chronic smoking for at least 1 year
* At least primary school graduate and can speak Turkish
* Having a smartphone and internet access
* No communication barrier (speech, vision or hearing problem)
* Individuals who agree to participate in the research.

Exclusion Criteria:

* Patients with positive CIS (carcinoma in situ)
* Patients with minimal invasion of the lamina propria and above
* Patients with extravesical extension
* Patients with synchronous and metachronous tumors
* Communication disability (speech, vision or hearing problem)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy for managing chronic disease 6-item scale. | Change from chronic disease self-efficacy at 12 months
  The scale is rated on a 10-point scale ranging from "not at all sure" to "very sure". The score obtained from the scale is the average of 6 items, and high scores indicate high self-efficacy. If more than one answer is given to an item and the items follow each other, the lower score is included in the calculation. In order to calculate the scale, at least 4 items must be answered. The Croncbach's alpha coefficient was 0.91 and the mean of the original scale was 5.17 ± 2.22. Turkish validity and reliability was done by İncirkuş and Nahcivan (2020). The Cronbach's alpha coefficient of the scale was found to be 0.90.
Glover Nilsson Smoking Behavioral Questionnaire | Change from smoking behavior at 12 months
  The Turkish validity and reliability of the scale was done by Sancar. The scale was created as a scale with 11 questions as a result of the Turkish adaptation study, and each question is scored from 0 to 4 with a 5-option scoring system. Behavioral addiction score below 12 is mild, 12 and 22 moderate, 23-33 strong, 33 above very strong behavioral addiction score has been suggested. The scale is a valid and reliable scale that can be used to determine the behavioral aspect of smoking addiction of smokers, both in its one-dimensional and 2-dimensional form. The Croncbach alpha coefficient was found to be 0.82. This value indicates that the scale is quite reliable in terms of internal consistency. The "Conditioning and Significance" sub-dimension of the scale consists of 5 items and the Cronbach's alpha coefficient is 0.762. The "Handling and Emotions" sub-dimension consists of 6 items and the Cronbach's alpha coefficient is 0.735.

SECONDARY OUTCOMES:
Tumor Recurrence | Change from tumor recurrence and progression at 12 months
  Tumor recurrence will be examined by cystoscopy at the 3rd and 12th months after the intervention.
Progression | Change from progression at 12 months
  Progression will be examined by cystoscopy at the 3rd and 12th months after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: İrem Nur Özdemir, PhD, RN, Principal Investigator — Bakırköy Dr. Sadi Konuk
Locations (1):
- İrem Nur Ozdemir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Spencer JC, Wheeler SB. A systematic review of Motivational Interviewing interventions in cancer patients and survivors. Patient Educ Couns. 2016 Jul;99(7):1099-1105. doi: 10.1016/j.pec.2016.02.003. Epub 2016 Feb 8. PMID 26879805
- [Result] Taylor KL, Williams RM, Li T, Luta G, Smith L, Davis KM, Stanton CA, Niaura R, Abrams D, Lobo T, Mandelblatt J, Jayasekera J, Meza R, Jeon J, Cao P, Anderson ED; Georgetown Lung Screening, Tobacco, and Health Trial. A Randomized Trial of Telephone-Based Smoking Cessation Treatment in the Lung Cancer Screening Setting. J Natl Cancer Inst. 2022 Oct 6;114(10):1410-1419. doi: 10.1093/jnci/djac127. PMID 35818122
- [Result] Wakefield M, Olver I, Whitford H, Rosenfeld E. Motivational interviewing as a smoking cessation intervention for patients with cancer: randomized controlled trial. Nurs Res. 2004 Nov-Dec;53(6):396-405. doi: 10.1097/00006199-200411000-00008. PMID 15586136
- [Result] Thomsen T, Tonnesen H, Okholm M, Kroman N, Maibom A, Sauerberg ML, Moller AM. Brief smoking cessation intervention in relation to breast cancer surgery: a randomized controlled trial. Nicotine Tob Res. 2010 Nov;12(11):1118-24. doi: 10.1093/ntr/ntq158. Epub 2010 Sep 20. PMID 20855414